CLINICAL TRIAL: NCT05571111
Title: A Randomised, Assessor-blind, Active-controlled, Parallel-group, Dose-finding Trial to Investigate the Efficacy and Safety of FE 999302 for Triggering of Final Follicular Maturation in Women Undergoing Controlled Ovarian Stimulation
Brief Title: Clinical Research Study to Learn About the Effect and Safety of Different Doses of FE 999302 When Given as a Single Dose for Final Development of the Eggs After Ovarian Stimulation
Acronym: TIFFANY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on company decision to close the project. No trial participants received any study drug.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000298
Record Dates: First submitted 2022-09-28; First posted 2022-10-07 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose 1 of FE 999302 (Experimental): Subcutaneous injection of Dose 1 of FE 999302 as a single dose.
  Interventions: Drug: FE 999302
- Dose 2 of FE 999302 (Experimental): Subcutaneous injection of Dose 2 of FE 999302 as a single dose.
  Interventions: Drug: FE 999302
- Dose 3 of FE 999302 (Experimental): Subcutaneous injection of Dose 3 of FE 999302 as a single dose.
  Interventions: Drug: FE 999302
- 250 μg OVITRELLE (Active Comparator): Subcutaneous injection of 250 μg of OVITRELLE. 0.5 mL as a single dose.
  Interventions: Drug: Ovitrelle
- 10,000 IU NOVAREL (Active Comparator): Subcutaneous injection of 10,000 IU NOVAREL.
  1 mL as a single dose.
  Interventions: Drug: Novarel

INTERVENTIONS:
Drug: FE 999302 — Subcutaneous injection as a single dose. 3 different doses
  Other Names: recombinant hCG
  Arms: Dose 1 of FE 999302; Dose 2 of FE 999302; Dose 3 of FE 999302
Drug: Ovitrelle — Subcutaneous injection as a single dose. 250 µg (0.5 mL)
  Arms: 250 μg OVITRELLE
Drug: Novarel — Subcutaneous injection as a single dose. 10,000 IU (1 mL)
  Arms: 10,000 IU NOVAREL

SUMMARY:
The primary purpose of this trial is to compare three different doses of FE 999302 with 250 µg OVITRELLE and 10,000 IU NOVAREL on oocyte maturity when administered as a single dose for final development of the oocytes in women undergoing controlled ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women between the ages of 18 and 42 years. The subjects must be at least 18 years (including the 18th birthday) and no more than 42 years (up to the day before the 43rd birthday) when they sign the informed consent.
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II or with partners diagnosed with male factor infertility, eligible for in vitro fertilisation (IVF) and/or intracytoplasmic sperm injection (ICSI) using fresh or frozen ejaculated sperm from male partner or sperm donor.
* Infertility for at least 1 year before screening for subjects <35 years or for at least 6 months for subjects ≥35 years (not applicable in case of tubal or severe male factor infertility).
* No more than two controlled ovarian stimulation cycles initiated, regardless outcome (taking exclusion criteria 3, 4, and 5 into account).
* Regular menstrual cycles of 24-35 days (both inclusive), presumed to be ovulatory.

Exclusion Criteria:

* Known polycystic ovary syndrome (PCOS) associated with anovulation or known endometriosis stage III-IV (American Society for Reproductive Medicine, 2012).
* Considered unsuitable for controlled ovarian stimulation with a starting dose of 150 or 225 IU/day highly purified human menopausal gonadotropin (HP-hMG), as judged by the investigator.
* Poor response in a previous controlled ovarian stimulation cycle using a gonadotropin starting dose of 150 IU/day or higher. Poor response is defined as <4 oocytes retrieved, or cycle cancellation prior to oocyte retrieval due to inadequate follicular development.
* Excessive ovarian response in a previous controlled ovarian stimulation cycle for IVF/ICSI using a daily FSH/hMG dose of ≤225 IU, defined as ≥25 oocytes retrieved or cycle cancellation prior to oocyte retrieval due to excessive ovarian response, including risk of ovarian hyperstimulation syndrome (OHSS).
* Severe OHSS in a previous controlled ovarian stimulation cycle.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Number of metaphase II (MII) oocytes | On the day of oocyte retrieval (2 days after triggering)

SECONDARY OUTCOMES:
Number of oocytes retrieved | On the day of oocyte retrieval (2 days after triggering)
Number of fertilised (2 pronuclei) oocytes | On day 1 insemination (3 days after triggering)
Number and quality of embryos on day 3 after oocyte retrieval | Day 3 after insemination (5 days after triggering)
Number and quality of blastocysts on day 5 after oocyte retrieval | Day 5 after insemination (7 days after triggering)
Serum hormone concentrations of progesterone | Blood samples for analysis of circulating concentrations of progesterone will be drawn at several visits from day of triggering up to 22 days after triggering
Serum hormone concentrations of 17-OH-progesterone | Blood samples for analysis of circulating concentrations of 17-OH-progesterone will be drawn at several visits from day of triggering up to 22 days after triggering
Serum hormone concentrations of estradiol | Blood samples for analysis of circulating concentrations of estradiol will be drawn at several visits from day of triggering up to 22 days after triggering
Serum hormone concentrations of follicle stimulating hormone (FSH) | Blood samples for analysis of circulating concentrations of follicle stimulating hormone (FSH) will be drawn at several visits from day of triggering up to 22 days after triggering
Serum hormone concentrations of luteinising hormone (LH) | Blood samples for analysis of circulating concentrations of luteinising hormone (LH) will be drawn at several visits from day of triggering up to 22 days after triggering
Positive βhCG (positive serum βhCG test 13-15 days after transfer) | 20-22 days after triggering
Clinical pregnancy (at least one gestational sac 5-6 weeks after transfer) | 6-7 weeks after triggering
Vital pregnancy (at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after transfer) | 6-7 weeks after triggering
Ongoing pregnancy (at least one intrauterine viable fetus 10-11 weeks after transfer) | 11-12 weeks after triggering
Serum hCG concentrations at end-of-stimulation, the day after triggering, at oocyte retrieval, on day 5 after oocyte retrieval (transfer), and on day 7-9 after oocyte retrieval (mid luteal phase) | Blood samples for analysis of circulating concentrations of hCG will be drawn at several visits from day of triggering up to 9-11 days after triggering
Ovarian hyperstimulation syndrome (OHSS), overall and by timing, grade, and severity | ≤9 days after triggering of final follicular maturation (early OHSS), >9 days after triggering of final follicular maturation (late OHSS)
  Early OHSS is defined as OHSS with onset ≤9 days after triggering of final follicular maturation. Late OHSS is defined as OHSS with onset >9 days after triggering of final follicular maturation.
Injection site reactions (redness, pain, itching, swelling, and bruising) assessed by the subject following administration of investigational medicinal product (IMP) | Immediately, 30 minutes, and 24 hours after injection
Treatment-induced anti-hCG antibodies, overall as well as with neutralising capacity | Day of triggering up until 19-28 days after triggering
Multi-fetal gestation | From day after blastocyst transfer (7 days after triggering) up until ongoing pregnancy (11-12 weeks after triggering)
Biochemical pregnancy | From day after blastocyst transfer (7 days after triggering) up until ongoing pregnancy (11-12 weeks after triggering)
Spontaneous abortion | From day after blastocyst transfer (7 days after triggering) up until ongoing pregnancy (11-12 weeks after triggering)
Ectopic pregnancy (with and without medical/surgical intervention) | From day after blastocyst transfer (7 days after triggering) up until ongoing pregnancy (11-12 weeks after triggering)
Vanishing twins | From day after blastocyst transfer (7 days after triggering) up until ongoing pregnancy (11-12 weeks after triggering)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (3):
- Spain (3):
  - Ferring Investigational Site, Madrid
  - Ferring Investigational Site, Seville
  - Ferring Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: No